CLINICAL TRIAL: NCT01636544
Title: Infectious Aetiology of Potentially Malignant Disorders and Squamous Cell Carcinomas of the Oral Cavity
Acronym: INECOC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Pasteur (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2011-45
Record Dates: First submitted 2012-07-06; First posted 2012-07-10 (Estimated); Last update posted 2022-04-26 (Actual); Status verified 2019-08

CONDITIONS: Squamous Cell Carcinoma of the Oral Cavity; Leukoplakia Oral
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Leukokeratosis, Hereditary Mucosal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- contralateral healthy tissue biopsy (Experimental)
  Interventions: Procedure: contralateral healthy tissue biopsy

INTERVENTIONS:
Procedure: contralateral healthy tissue biopsy — At the time of surgery, a part of the specimen, plus a biopsy of the healthy (control) contralateral mucosa (i.e. right border of the tongue for a SCC of the left border, left cheek for a dysplasia of the right cheek and so on) will be harvested for research and immediately frozen at -80°C first in dry ice, then in a -80°C freezer.

SUMMARY:
Recent studies estimated that 15 to 20% of all cancers in humans are associated with viruses. Among oral cancer about 90% are oral squamous cell carcinomas (OSCC). Alcohol and tobacco consumption have been recognized for years as the main risk factors for development of OSCCs. However, 10 to 20% of patients suffering from OSCCs are non-smokers and/ or non-drinkers. Consequently, the hypothesis of another agent responsible has risen. Indeed, several studies have suggested the possibility that a virus could be associated with or be a causal agent of OSCC. The first objective is to detect and characterize the presence of infectious agent (mostly virus) transcripts in pre-malignant or malignant tumours from patients with OSCCs.The secondary objectives are (i) to associate and (ii) if possible define a causality link between these agents and a subset of potentially malignant disorders and/or OSCCs.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years,
* For subgroup "potentially malignant disorder : clinical diagnosis of leukoplakia,
* For subgroup "OSCC" : histological diagnosis of OSCC,
* Patient who never smoked, or light smoker, (≤5 pack-year) or 15 years of cessation,
* Patient who never drank, or light drinker (≤ 20 g/day for men and 10g/day for women) or 15 years of cessation,
* Informed consent signed.

Exclusion Criteria:

• Previous treatment of oral cancer,

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2012-06-15 (Actual); Primary Completion 2015-12-10 (Actual); Study Completion 2016-01-31 (Actual)

PRIMARY OUTCOMES:
Detection and characterization of HPV (human papillomavirus)by using qPCR (quantitative polymerase chain reaction) method. | 30 months
  qPCR method
Detection of others infectious agents | 30 months
  (i) a high -density panviral resequencing microarray (RMA) and (ii) High-Throughput Sequencing (HTS)

SECONDARY OUTCOMES:
Clonality of viral agent | 30 months
  RMA and HTS

CONTACTS AND LOCATIONS:
Overall Officials: Chloé Bertolus, MD, Principal Investigator — APHP; Antoine Gessain, PhD, Study Chair — Institut Pasteur
Locations (1):
- hôpital la Pitié Salpêtrière - APHP, Paris, France